CLINICAL TRIAL: NCT00556231
Title: Use of Multi-site Near Infrared Spectroscopy (NIRS) Monitoring for Global Hemodynamic Assessment During Exercise Testing in Children With and Without Heart Disease
Brief Title: Multi-site Near Infrared Spectroscopy (NIRS) Monitoring of Children During Exercise
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, John Hambrook, Assistant Professor, Pediatrics, Cardiology, Medical College of Wisconsin
Other Study IDs: CHW 07/198
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Congenital Heart Disease
Keywords: NIRS; cardiac output; anaerobic threshold; exercise stress; congenital heart defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Children with congenital heart lesions - males/females, ages 6-20, scheduled for a regular stress test
- 2: Children without congenital heart lesions - males/females, ages 6-20, scheduled for a regular stress test
- 3
- 4
- 5
- 6

SUMMARY:
Near Infrared Spectroscopy (NIRS) monitoring has proven beneficial in increasing safety and improving patient care during pediatric cardiac surgery and during Pediatric Intensive Care Unit (PICU) stays. NIRS estimates the amount of oxygen in tissues by comparing the tissue's absorption of two wavelengths of light corresponding to hemoglobin carrying oxygen and hemoglobin without oxygen.

During cardiac surgery, multi-site NIRS monitoring is used to determine the heart's output by comparing the amount of oxygen available to discrete regions of the body nourished by different parts of the circulatory system. NIRS leads placed on the forehead detect oxygen available to the brain (cerebral), while leads placed over the kidney reflect oxygen available to the internal organs (somatic).

NIRS monitoring has been used for studying muscle oxygen usage during exercise in normal and disease states. Cerebral oxygenation at peak exercise at has been studied with NIRS monitoring. The use of multi-site NIRS monitoring during exercise stress testing for studying cardiac output through the patterning of somatic and cerebral oxygenation in combination with exercise stress test data has not been researched.

We hypothesize that addition of multi-site NIRS monitoring to the standard data collection already achieved during exercise testing, will enable calculation of anaerobic threshold and cardiac output prediction. This will assist in determining appropriate timing for surgical intervention, predicting the post operative course and testing response to medication.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents from age 6 to 20 undergoing exercise stress testing on treadmill

Exclusion Criteria:

* Children and adolescents unable to exercise or unable to follow directions or unable to understand English.

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents from age 6 to 20 undergoing exercise stress testing
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
regional oxygen saturations in 4 sites | during exercise stress testing

CONTACTS AND LOCATIONS:
Overall Officials: John Hambrook, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Result] Danduran MJ, Dixon JE, Rao RP. Near infrared spectroscopy describes physiologic payback associated with excess postexercise oxygen consumption in healthy controls and children with complex congenital heart disease. Pediatr Cardiol. 2012 Jan;33(1):95-102. doi: 10.1007/s00246-011-0097-3. Epub 2011 Sep 3. PMID 21892649
- [Result] Rao RP, Danduran MJ, Loomba RS, Dixon JE, Hoffman GM. Near-infrared spectroscopic monitoring during cardiopulmonary exercise testing detects anaerobic threshold. Pediatr Cardiol. 2012 Jun;33(5):791-6. doi: 10.1007/s00246-012-0217-8. Epub 2012 Feb 19. PMID 22349729
- [Derived] Rao RP, Danduran MJ, Hoffman GM, Ghanayem NS, Berger S, Frommelt PC. Cerebral hemodynamics in the presence of decreased systemic venous compliance in patients with Fontan physiology may limit anaerobic exercise capacity. Pediatr Cardiol. 2010 Feb;31(2):208-14. doi: 10.1007/s00246-009-9585-0. PMID 19915888